CLINICAL TRIAL: NCT01694472
Title: Phase 1 Study of MAGE-A4 TCR Gene-Modified T Cells to Treat Malignant Tumors
Brief Title: Clinical Safety and Preliminary Efficacy of MAGE-A4 TCR Gene-Modified T Cells to Treat Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIH-RXB-201205002
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-09

CONDITIONS: Malignant Solid Tumors

ARMS (1):
- MAGE-A4 TCR Gene-Modified T Cells (Experimental)
  Interventions: Biological: MAGE-A4 TCR Gene-Modified T Cells

INTERVENTIONS:
Biological: MAGE-A4 TCR Gene-Modified T Cells — The study consists of a 2-dose escalation scheme, and the patient receives twice in each dose. The starting dose is 1-3 x 10^9 cells of each TCR gene-modified cells and the second one is 3-8 x 10^9 cells of each TCR gene-modified cells. Two weeks after the first infusion the patient receives the same dose again, followed by infusions of IL-2 for 5 days. Thereafter, the patient receives peptide vaccinations on days 21 and 28.

SUMMARY:
The purpose of this study is to evaluate the clinical safety and preliminary efficacy of MAGE-A4 TCR Gene-Modified T lymphocytes in the treatment of malignant solid tumor patients, such as malignant melanoma and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male or female
* Age: from 18 to 80 years
* Patients must have histologically confirmed solid tumors that have failed standard therapies (surgery, chemotherapy, radiotherapy) and for which no curative options exist, including, but not limited to:

Non-Small Cell Lung Carcinoma Malignant melanoma Esophageal carcinoma Head and neck carcinoma

* HLA-A*24:02
* MAGE-A4 positive in the test by RT-PCR on tumor tissue or immunohistochemistry of resected tissue of the patient.
* PS ECOG 0 or <2
* Laboratory tests results 7 days before the start of treatment:

White blood cells: more than 3.0 × 109/L Platelets: more than 100 × 109/L Neutrophils: more than 1.5 × 109/L Hemoglobin: more than 80g/L Serum glutamate pyruvate transaminase: less than 2.5 folds of the upper normal limit (ULN) Serum glutamic-oxal (o) acetic transaminase: less than 2.5 × ULN Serum bilirubin: less than 1.25 × ULN Serum creatinine: less than 1.25 × ULN

* Pregnancy test: the test of women of child-bearing period must be negative 7 days before the start of treatment
* Contraception: male and female subjects of child-bearing period must adopt a reliable method of contraception before entry into this study until 30 days after stopping this study
* Informed consent: subject must have the ability to understand and voluntarily sign a written informed consent

Exclusion Criteria:

* Patients with life-threatening condition or complication other than their basic disease
* Pregnant or lactation. Patients both males and female with reproductive potential (i.e. menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration
* Active systemic infections
* History of neoplasms: other neoplasms
* Medical history: active CNS disease, or congestive heart failure, or severe coronary artery disease, or cardiac arrhythmias, or concomitant corticosteroid therapy
* Metastasis: clinical symptoms of brain metastasis
* Other clinical trial: the subject received other clinical trial before this study
* Laboratory tests: the serum test of human immunodeficiency virus, or hepatitis B virus, or hepatitis C virus was positive
* Compliance: poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 12 months
  CR + PR = ORR

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China